CLINICAL TRIAL: NCT03974815
Title: Augmentative Transcranial Direct Current Stimulation (tDCS) in Patients With Bipolar Depression: RCT, IIT Study.
Brief Title: tDCS(Transcranial Direct Current Stimulation) Efficacy in Bipolar Depression : RCT Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ybrain Inc. (Industry)
Responsible Party: Principal Investigator, Woojae Myung, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YB_ST_IIT1901
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: tDCS
Keywords: tDCS; Bipolar disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Active stimulation group: 2mA, 30min (1min ramping up/down) Sham stimulation group: 0mA, 30min (1min ramping up/down)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVE (Experimental): Active stimulation (tDCS) will be used in the dose of 2mA /30 min per day, for 6weeks. (minimum 5 times per week)(total of 30~42 sessions)
  Interventions: Device: ACTIVE
- SHAM (Sham Comparator): Sham stimulation (tDCS) will be used in the dose of 0mA /30 min per day, for 6weeks. (minimum 5 times per week)(total of 30~42 sessions)
  Interventions: Device: SHAM

INTERVENTIONS:
Device: ACTIVE — We will use 28.26cm^2 round electrodes and a 2mA current for 30 minutes per day. This montage is known as "bifrontal" setup(F3-Anode, F4-Cathode) and has been previously used in major depression trials.
  Arms: ACTIVE
Device: SHAM — We will use 28.26cm^2 round electrodes and a 0mA current for 30 minutes per day. This montage is known as "bifrontal" setup(F3-Anode, F4-Cathode) and has been previously used in major depression trials.
  Arms: SHAM

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation (tDCS) is effective and safe in the treatment Bipolar depression.

Randomized, double-blind Controlled Clinical Trial. Subjects Adults (between 19 and 65 years of age) with Bipolar depression who meet the inclusion criteria and who agree to participate in the study Will recruit from clinical referrals.

* Active tDCS Anode - left DLPFC Cathode - right DLPFC Electric current is 2mA - Current is applied for 30 min
* Sham tDCS Same assembly is used Current is applied for 1 min

Both groups 30~42 stimulation sessions on consecutive days.

Baseline(visit 1), 2 week(visit 2), 4 week(visit 3), 6 week(visit 4), and 12 week(visit 5) Check compliance with mobile application(MINDD-CONNECT) connections.

DETAILED DESCRIPTION:
Assessment:

Depression rating scale: HAM-D(Hamiltion Depresiion Rating Scale), HAM-A(Hamilton Anxiety Rating Scale) Maniac rating scale: YMRS(Young Mania rating scale) CGI-BP(Clinical Global Impression-Bipolar) Q-LES-Q-SF(Quality of Life Enjoyment and Satisfaction Short form) Q-LES-Q-Q(Quality of Life Enjoyment and Satisfaction Questionnaire) qEEG(Quantitative Electroencephalography)

Check compliance with mobile application(MINDD-CONNECT) connections.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II of bipolar disorder meets the current major depression diagnostic criteria in DSM-5
* CGI Severity of lightness score ≥ 4 points
* Taking mood stabilizers for at least four weeks before the day of screening

Exclusion Criteria:

* A history of clinically significant internal neurological disorders or head injury
* mental retardation or cognitive impairment that will affect to make a consent form.
* Patients at risk of suicide that may require hospitalization as determined by clinicians
* A person who is determined to be excluded for using tDCS medical device for other reason (e.g. metal plate is inserted on head, etc.)
* A person who is determined to have problems with scalp deformation, inflammatory response or brain wave and attachment of direct current because of other dermatological problem
* A woman who disagree with medically allowed contraception* until 24 weeks after the application of investigational device among woman subject who is possible to get pregnant

  * Medically allowed contraception: condom, oral contraception for at least 3 month, injection or insert contraception, Intrauterine Device, etc.
* pregnant woman or lactating woman
* A person who is not suitable for this clinical trial based on principal investigator's determination other than above reasons

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
The changes in HAM-D | baseline, 2week, 4week, 6week
  The changes in HAM-D(Hamilton Depression scale) will constitute the major research outcome measure.
  HAM-D17
  * clinician-administered scale
  * assesses 17 items related to major depression (MD)
  * Individual items scored on 3 point (0 to 2) or 5 point scale (0 to 4)
    ; 0=absent, 4=most severe.
  * Total score: 0 to 66.
Response rate of treatment | baseline, 6week
  Response group: Reduce of HAM-D 50%

SECONDARY OUTCOMES:
HAM-A | baseline, 2week, 4week, 6week
  Hamilton Anxiety Rating Scale
  * Rating clinician-related
  * Main purpose to assess the severity of symptoms of anxiety
  * Population adults, adolescents and children
  * The scale consists of 14 items
  * Each item is scored on a scale of 0-4, with a total score range of 0-56
  * <17: mild severity, 18-24: mild to moderate severity, 25-30: moderate to severe
YMRS | baseline, 2week, 4week, 6week
  Young Mania Rating Scale
  * Rating clinician-related or other trained rater
  * Main purpose to assess the severity of symptoms of manic
  * Population young adults and children
  * The scale consists of 11 items
  * Each item is scored on a scale of 0-8 or 0-4, with a total score range of 0-60
  * The higher score, the worse it means.
CGI-BP | baseline, 2week, 4week, 6week
  Clinical Global Impression- Bipolar
Q-LES-Q-SF | baseline, 2week, 4week, 6week
  Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form

OTHER OUTCOMES:
qEEG | baseline, 2week
  The changes of qEEG analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Boondang Hospital, Seongnam-si, Boondang, Gyunggi, South Korea

REFERENCES:
- [Derived] Lee J, Lee CW, Jang Y, You JS, Park YS, Ji E, Yu H, Oh S, Ryoo HA, Cho N, Park JY, Yoon J, Baek JH, Park HY, Ha TH, Myung W. Efficacy and safety of daily home-based transcranial direct current stimulation as adjunct treatment for bipolar depressive episodes: Double-blind sham-controlled randomized clinical trial. Front Psychiatry. 2022 Sep 20;13:969199. doi: 10.3389/fpsyt.2022.969199. eCollection 2022. PMID 36203828